CLINICAL TRIAL: NCT05331612
Title: Blended Treatment for Problem Gambling and Gambling Disorder Combining Group Sessions and Online Modules: A Pilot Randomized Controlled Trial
Brief Title: Blended Treatment for Problem Gambling and Gambling Disorder Combining Group Sessions and Online Modules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARAMENI/189
Record Dates: First submitted 2022-03-01; First posted 2022-04-15 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Gambling Disorder; Problem Gambling
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blended intervention condition (Experimental): Blended intervention condition, consisting of 5 face-to-face group sessions lasting 2 hours every 2 weeks, alternated with the online treatment protocol carried out by the participants in a self-applied. The intervention has a period of duration of 13 weeks and it is composed by 8 modules (Motivation for change, Psychoeducation, Stimulus control, Cognitive restructuring, Urge surfing and emotion regulation, Planning of significant activities, Coping skills and exposure with response prevention, and Relapse prevention). These modules is based in the online platform and manualized protocol treatment "Sin jugar, ganas" (Díaz-Sanahuja et al., 2021).
  Interventions: Behavioral: Blended intervention condition
- Waiting list control condition (No Intervention): Waiting list control group receives the blended treatment when the intervention has finished in the experimental group (blended group intervention).

INTERVENTIONS:
Behavioral: Blended intervention condition — Participants receive the online protocol treatment and face-to-face sessions during 13 weeks.
  Other Names: BI
  Arms: Blended intervention condition

SUMMARY:
The main objective of present project is assess the preliminary efficacy of a blended psychological intervention, by comparing the improvements in the CBT and waiting list control groups of an evidence-based treatment protocol for problems related to gambling applied in a blended format (sessions through an online protocol treatment combining with face-to-face group sessions), as well as to evaluate the opinion and acceptance of the intervention.

DETAILED DESCRIPTION:
Gambling disorder and problem gambling are considered a public health problem around the world, not only because of the high costs of the treatments that it entails, otherwise by the increase in the numbers of young people who easily fall into gambling behavior and who can hardly leave problems with games of chance on their own.

The review of the scientific literature has shown that CBT is the psychological therapy that has shown the greatest scientific evidence and rigor over the years in the treatment of gambling disorder and problem gambling. In addition, the application of Information and Communication Technologies (ICTs), together with the characteristics of accessibility, immediacy and cost reduction, which show, has made it possible to carry out effective Internet-delivered Interventions. If investigators take into account the high rates of drop outs and the low adherence to treatment that exists among patients with behavioral addictions, as well as the current barriers encountered by patients, such as stigma, the costs of the sessions and the distance geographical location.

A new alternative and innovative treatment are blended interventions, although their research is still limited, their efficiency and effectiveness have been proven for the treatment of emotional disorders and substance addictions, such as smoking cessation. In the same way, the benefits which offers CBT group therapy are improvement the self-esteem, encourages problem solving and communication skills and mutual support.

Therefore, the objective of the present project will be to evaluate whether a blended intervention (group sessions plus Internet-based modules) for problem gambling and gambling disorder could lead to improved gambling outcomes compared to a waiting list control condition.The minimum number of participants diagnosed with gambling disorder and problem gambling, which will be randomly assigned to each of the two conditions, will be 30 participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Being able to understand, read and write Spanish.
* Having a computer and daily access to the Internet at home.
* Meeting criteria for gambling disorder or problem gambling according to the parameters established by the Norc Diagnostic Screening for gambling disorders (NODS) (Becoña, 2004),
* Availability and willingness to provide information about gambling behavior in the follow-ups.

Exclusion Criteria:

* Having any serious mental disorder.
* If the behavior comes to maniac from a maniac episode or from taking antidepressants
* Being high risk of suicide,
* Moderate or severe alcohol and substance use disorder according to the Mini International Neuropsychiatric Interview (MINI) (Sheehan et al.,1998).
* Any medical illness that conditions receiving treatment receives.
* Increasing in the dose of pharmacological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Gambling Symptom Assessment Scale (Kim et al., 2009). At baseline, post-module, post-treatment, 3, 6 and 12 months follow-up. | Up to 12 months.
  The G-SAS is a 12-item self-rated scale designed to assess gambling symptom severity and change during treatment. All items are scored on a 4-point scale, and the score ranges from 0 to 48: extreme=41-48, severe=31-40, moderate=21-30 and mild=8-20. The scale shows a higher internal consistency (α = 0.82).
Gambling-related cognitions scale (Del Prete et al., 2017). At baseline, post-treatment, 3, 6 and 12 months follow-ups. | Up to 12 months.
  The GRCS is a self-report which assessed the gambling cognitions through 23 items divided into 5 dimensions that are rated on a 7-point Likert-type scale (1 = I strongly disagree; 7 = I strongly agree). The reliability of each of the dimensions is adequate ID (α = 0.79), in adequate EJ (α = 0.72), in adequate CI (α = 0.7), in adequate PC (α = 0.73) and in good SI (α = 0.8). The degree of internal consistency of the total score of the scale was better (α = 0.9).

SECONDARY OUTCOMES:
Gambling Self-Efficacy Questionnaire (Winfree et al., 2013). At post-treatment, 3,6 and 12 months follow-ups. | Up to 12 months.
  The GSEQ is a self-report measure to assess an individual's perceived self-efficacy to control his or her gambling behavior in a variety of situations through 16 six-point Likert scale items. The total score is calculated through the average response given among all the items on the scale, ranging from 0 to 100. Higher scores denote greater confidence in the gambling behavior by the patient. It has shown a good internal consistency of .96.
The University of Rhode Island Change Assessment Scale (Gómez-Peña et al., 2011). At baseline, post-treatment, 3, 6 and 12 follow-ups. | Up to 12 months.
  The URICA is a self-report measure that includes 4 subscales measuring the stages of change of Prochaska & DiClemente (Pre-contemplation, Contemplation, Action, and Maintenance) (there is also a 24-item version) through 32 ítems. Responses are given on a 5-point Likert scale ranging from (1=strong disagreement to 5=strong agreement) (McConnaughy et al.,1983).The scores of each of the subscales range from 8 to 40, they are obtained through the five items that make up each of these. It shows internal consistency of .74.

CONTACTS AND LOCATIONS:
Overall Officials: Juana Bretón López, Professor, Study Director — University Jaume I
Locations (1):
- University Jaume I, Castellon, Castelló, Spain